CLINICAL TRIAL: NCT05975125
Title: The Effect of Vitamin C for Iron Supplementation During Pregnancy with Risk of Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 118/2566
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-06

CONDITIONS: Vitamin C Anemia; Pregnancy Anemia
Keywords: Vitamin C, Pregnancy with anemia
MeSH Terms: interventions — Ascorbic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron supplement with Vitamin C (Experimental): Vitamin C with Iron supplement
  Drug:
  Vitamin C 500mg Triferdine(Component: Iodine 0.15 mg, Iron 60.81 mg, Folic acid 0.4 mg)
  Interventions: Drug: Vitamin C 500 MG Oral Tablet
- Iron supplementation alone (No Intervention): Iron supplement alone Drug: Triferdine Component: Iodine 0.15 mg, Iron 60.81 mg, Folic acid 0.4 mg

INTERVENTIONS:
Drug: Vitamin C 500 MG Oral Tablet — compare between Vitamin C with iron supplement and iron supplement alone in prevention of anemia in pregnancy.
  Arms: Iron supplement with Vitamin C

SUMMARY:
Anemia is a common problem during pregnancy. Most studies have demonstrated that anemia during pregnancy have adverse effects on their pregnancy outcome, which is important and should pay attention to prevent and solve such problems. The most common cause of anemia is iron deficiency. Several studies reveal that Vitamin C promotes iron absorption. In this study we will compare between Vitamin C with iron supplement and iron supplement alone in prevention of anemia in pregnancy.

DETAILED DESCRIPTION:
Anemia in pregnancy associated with Diabetes during pregnancy 15.9 % Fetal abnormalities in blood oxygen causing fetal non reassuring 9.4% , Preterm delivery 8.2 %, Amniotic fluid insufficiency 1.95 %, 10.6 % of infants had complications after birth, 9.7 % of infants were hospitalized in intensive care units with birth weight less than 2,500 grams . (Low birth weight) 4.9%, anemia also significantly increased the likelihood of blood transfusion during pregnancy.

There is also a study on the risk of developing anemia such as more than 2 pregnancies, Teenage pregnancy, Advanced maternal age more than 35 years old, Mothers with a body mass index below 18 are at increased risk of developing anemia. The most common cause of anemia during pregnancy is iron deficiency. This may be caused by receiving the element. not enough iron or there is a loss of iron from blood loss which is important and should pay attention to prevent and solve such problems. Which Vitamin C promotes iron absorption. Vitamin C combined with iron has been studied. It clearly increases hemoglobin and hematocrit. And is safe for pregnant women and babies. There is also no evidence that vitamin C is a carcinogen, or a cause of birth defects or toxicity. However, there are no studies related to the combination of vitamin C and iron in pregnant women at risk of anemia. To solve the problem and prevent the consequences of the above mentioned anemia. In this study we will compare between Vitamin C with iron supplement and iron supplement alone in prevention of anemia in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman Antenatal care at Rajavithi Hospital
2. Singleton pregnancy
3. Provide inform consent with both patient and her husband
4. Gestational age between 14-28 weeks
5. Risk of anemia during pregnancy, including more than 2 pregnancies, teenage pregnancy, advanced maternal age over 35 years old, mothers with body mass index below 18.

5. Pregnant women with hemoglobin greater than 10.5 g/dL, hematocrit greater than 32 % in the first antenatal blood results. 6. Giving birth at Rajavithi Hospital 7. Can communicate and understand Thai language very well

Exclusion Criteria:

1. Receive vitamin C supplements during the program
2. HIV infection
3. Iron deficiency anemia or blood diseases such as thalassemia
4. Gastrointestinal bleeding
5. Antenatal hemorrhage
6. Allergic to vitamin C or iron
7. Congenital diseases including kidney disease, liver disease, joint disease and bleeding disorders.
8. Symptoms that indicate infection, such as fever, sore throat, sputum, diarrhea, loose stools, etc.
9. History of iron intake within the past 3 months
10. Received blood components within the past 3 months or while participating in a research project
11. Giving birth during the drug trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant woman
Enrollment: 100 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
To compare hemoglobin and hematocrit levels | 2 months after intervention
  To compare hemoglobin and hematocrit levels between groups receiving vitamin C with iron and the group receiving only iron supplement

SECONDARY OUTCOMES:
maternal and fetal pregnancy outcomes | after intervention until delivery
  To compare maternal and fetal pregnancy outcomes such as postpartum haemorrhage, blood transfusion after birth, birth body weight, gestational age at childbirth, the health of the baby after birth, etc., among the groups that received vitamin C and iron intake compare with the group that received only iron supplement alone.
ratio of vitamin C | 2 months after intervention
  To study the ratio of vitamin C and iron supplement in prevention of anemia in pregnancy.
side effects after receiving vitamin C | 2 months after intervention
  To study the side effects after receiving vitamin C during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi, Phaya Thai, ratchathewi, Thailand